CLINICAL TRIAL: NCT01926860
Title: Immune Response to Pneumococcal Conjugate Vaccine in Adults Receiving Hepatitis a Vaccine At the Same Time
Brief Title: PCV13 + Hepatitis a Vaccine for Adults
Acronym: PCV13+HepA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anu Kantele, Associate Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PCV13 adults + Hep A
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Measurement of Immune Response to Prevenar13; Measurement of Immune Response to Hepatitis a
Keywords: Prevenar13; pneumococcal conjugate vaccine; Epaxal; hepatitis A vaccine
MeSH Terms: conditions — Hepatitis | interventions — 13-valent pneumococcal vaccine; Hepatitis A Vaccines; epaxal berna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study group - Prevenar®13 and Hepatitis A vaccines (Experimental): Study group (group 1) - Prevenar®13 and Hepatitis A: one dose of each vaccine administered on Day 0
  Interventions: Biological: Prevenar13; Biological: Hepatitis A vaccine
- Pneumococcal conjugate vaccine -Control group - Prevenar®13 (Active Comparator): PCV -Control group (group 2) - Prevenar®13: one vaccine injection administered on Day 0
  Interventions: Biological: Prevenar13
- HepA -Control group - Hepatitis A vaccine (Active Comparator): HepA -Control group (group 3) - Hepatitis A vaccine: one vaccine injection administered on Day 0
  Interventions: Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: Prevenar13
  Arms: Pneumococcal conjugate vaccine -Control group - Prevenar®13; Study group - Prevenar®13 and Hepatitis A vaccines
Biological: Hepatitis A vaccine
  Other Names: Epaxal
  Arms: HepA -Control group - Hepatitis A vaccine; Study group - Prevenar®13 and Hepatitis A vaccines

SUMMARY:
The present study explores whether a simultaneously given hepatitis A vaccine (Epaxal) will have an impact on the immune response to PCV13 (pneumococcal conjugate vaccine; Prevenar13) vaccine in adults. The immune response to PCV13 is measured as levels of serotype specific serum antibodies and their opsonophagocytic activity. The results of volunteers receiving PCV13 and Epaxal will be compared to that in a control groups of adults receiving either hepatitis A or PCV13 vaccines only.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥50
2. General good health as established by medical history and physical examination
3. Written informed consent
4. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable.
5. Available for all visits scheduled in this study.
6. No previous Pnc vaccination
7. No previous hepatitis A vaccine
8. No other vaccines administered 30 days prior to or during the study

Exclusion Criteria:

1. Previous pneumococcal or hepatitis A vaccination
2. Immunization with any other vaccine (oral or parenteral) within 4 weeks prior to study start or planned vaccination during the study
3. Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of vaccine; patients using oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent are excluded; inhaled or topical steroids are allowed
4. Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
5. Pregnancy or lactation
6. Acute disease at the time of enrollment (defined as the presence of a moderate or severe illness with or without fever (fever is defined as body temperature of ≥38 °C).
7. Alcohol or drug abuse
8. Suspected non-compliance
9. Use of any investigational drug within 30 days preceding the study vaccine, or planned use during the study period
10. Any clinically significant history of known or suspected anaphylaxis or hypersensitivity reaction based on the judgement of the investigator
11. Employee at the investigational site, relative or spouse of the investigator
12. Any other criteria which, in the investigator's opinion, would compromise the ability of the subject to participate in the study, the subject's well-being, or the outcome of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2013-08-24 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Immune response to PCV13 | 2 years
  - To study whether a simultaneously given hepatitis A vaccine (Epaxal) will have an impact on the immune response to PCV13 (Prevenar13) vaccine in adults. The immune response to PCV13 is measured as levels of serotype specific serum antibodies and their opsonophagocytic activity. The results of volunteers receiving PCV13 and Epaxal will be compared to that in a control group of adults receiving PCV13 vaccine only.

SECONDARY OUTCOMES:
Immune response to Hep A vaccine | 2 years
  - To study whether a simultaneously given PCV13 vaccine will have an impact on the immune response to hepatitis A vaccine in adults. The immune response to hepatitis A vaccine is measured as levels of serum antibodies (ELISA). The results of volunteers receiving PCV13 and hepatitis A will be compared to that in a control group of adults receiving hepatitis A vaccine only.

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, Assoc. prof., Principal Investigator — Helsinki University Central Hospital; Lars Rombo, Professor, Principal Investigator — Sörmland County Council, Centre for Clinical Research
Locations (2):
- Aava Medical Centre, Helsinki, Finland
- Department of Infectious Diseases, Eskilstuna, Sweden

REFERENCES:
- [Background] Riekkinen M, Pakkanen SH, Hutse V, Roukaerts I, Ollgren J, Kayhty H, Herzog C, Rombo L, Kantele A. Coadministered pneumococcal conjugate vaccine decreases immune response to hepatitis A vaccine: a randomized controlled trial. Clin Microbiol Infect. 2023 Dec;29(12):1553-1560. doi: 10.1016/j.cmi.2023.08.006. Epub 2023 Aug 10. PMID 37572831